CLINICAL TRIAL: NCT03023696
Title: A Randomized, Prospective Study Determining the Impact of Prophylactic Bilateral Foraminotomy During Cervical Decompression on C5 Palsy
Brief Title: Can Prophylactic Foraminotomy Prevent C5 Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Thomas Mroz, MD, Institute Chair, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-353
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Myelopathy, Compressive; Radiculopathy, Cervical; C5 Palsy
Keywords: C5 Palsy; foraminotomy
MeSH Terms: conditions — Spinal Cord Compression; Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foraminotomy Group (Experimental): Prophylactic bilateral cervical keyhole foraminotomy will be done in addition to their decompression surgery
  Interventions: Procedure: Bilateral Cervical Keyhole Foraminotomy; Procedure: Cervical Decompression
- Control Group (Active Comparator): Cervical decompression will be done without prophylactic bilateral foraminotomy
  Interventions: Procedure: Cervical Decompression

INTERVENTIONS:
Procedure: Bilateral Cervical Keyhole Foraminotomy — Under microscopic or loop magnification, a high-speed burr is used to perform the foraminotomy. The keyhole foraminotomy begins at the lamina-facet junction, with careful consideration of the amount of facet resection. Typically, only the medial one third is drilled. Then a 1- or 2-mm Kerrison punch can be carefully placed over the nerve root and then used to undercut the facet, ensuring that the spine is not destabilized by the foraminotomy. The amount of facet resection must not exceed 50% in order to preserve spine stability.
  Arms: Foraminotomy Group
Procedure: Cervical Decompression — Cervical decompression for myelopathy, including the following procedures: laminoplasty, laminectomy, discectomy and fusion

SUMMARY:
C5 palsy (C5P) is a well-known, although rare complication of cervical spine decompression surgery. In severe forms, C5P causes debilitating upper extremity weakness involving the deltoids and/or biceps brachii muscles, ultimately diminishing these patients' quality of life. Furthermore, about half of patients with C5P present with sensory deficits and/or intractable pain in addition to the muscle weakness.

Prophylactic bilateral foraminotomy at the C5 level during cervical decompression surgery has been studied recently with the hope that it will minimize the risk of developing a C5 nerve root palsy postoperatively. Although the current literature provides some support for this claim, there are insufficient data establishing this technique as a proven measure to reduce the incidence of C5P. In the present study, we seek to evaluate the effect of bilateral foraminotomy on postoperative C5P incidence rates.

Bilateral foraminotomy has been correlated with a reduced risk of developing C5P following cervical decompression surgery, but an identical foraminotomy procedure has never been applied in a randomized manner to all qualifying patients in a study. Additionally, prophylactic foraminotomy has only been prospectively studied during laminoplasty. In the proposed study, bilateral foraminotomy will be randomized to patients receiving cervical decompression surgery (laminoplasty, laminectomy, fusion). This is a multicenter randomized trial, including the following sites: Cleveland Clinic, Columbia University Medical Center, and University of Southern California Spine Center. Patients undergoing cervical decompression surgery will be consented and enrolled if they meet the inclusion and exclusion criteria. Subsequently, incidence of C5P will be monitored to determine efficacy of prophylactic C5 bilateral foraminotomy during cervical decompression.

DETAILED DESCRIPTION:
Introduction:

C5 palsy (C5P) is a well-known, although rare complication of cervical spine decompression surgery.1,2 In severe forms, C5P causes debilitating upper extremity weakness involving the deltoids and/or biceps brachii muscles, ultimately diminishing these patients' quality of life.3 Furthermore, about half of patients with C5P present with sensory deficits and/or intractable pain in addition to the muscle weakness.5 Fortunately, almost all cases of C5P present unilaterally. The deficit is typically quantified and diagnosed using each patient's manual muscle test (MMT) score (rating 0-5). The American Medical Association impairment rating guide grades the MMT as follows: Grade 0 = no perceptible muscle contraction; Grade 1 = muscle contraction palpable, but no motion; Grade 2 = motion of the part only with gravity reduced; Grade 3 = muscle can hold the part in the test position against gravity alone; Grade 4 = patient can move the part through the full range of active motion against "some" resistance; Grade 5 = patient can move the part through the full active range of motion against "full" resistance. C5P is defined as: a reduction of at least 1 in deltoid and/or biceps brachii scores compared to preoperative scores, without any deterioration of myelopathic symptoms.5

Although a uniform understanding of the etiology and mechanism of C5P is not yet established, certain hypotheses have gained recognition. One prominent hypothesis, called the tethering phenomenon, suggests that following decompression, posterior shift of the cord produces traction on the nerve root resulting in a nerve root lesion. Other, less agreed upon hypotheses include: inadvertent injury to the nerve root during surgery, spinal cord ischemia, segmental spinal cord disorder, and reperfusion injury of the spinal cord. As the pathogenesis of C5P is uncovered, concerted efforts to minimize the incidence of this unfortunate complication have been undertaken.5

Prophylactic bilateral foraminotomy at the C5 level during cervical decompression surgery has been studied recently with the hope that it will minimize the risk of developing a C5 nerve root palsy postoperatively.6,7,8 Although the current literature provides some support for this claim, there are insufficient data establishing this technique as a proven measure to reduce the incidence of C5P. In the present study, we seek to evaluate the effect of bilateral foraminotomy on postoperative C5P incidence rates.

Background:

Komagata et al.7 performed a retrospective study to investigate preoperative risk factors that may cause postoperative C5P. The study included 305 cases of cervical expansive laminoplasty performed for spondylotic myelopathy or ossification of the posterior longitudinal ligament. No specific risk factors were found to be associated with higher incidence of C5P. However, bilateral partial foraminotomy was found to be effective in preventing C5P, with C5P occurring in 1 gutter (0.6%) in the foraminotomy group and in 12 gutters (4.0%) in the non-foraminotomy group (p<0.05).

Interestingly, preoperative anatomical measurements have been suggested to correlate with risk of developing C5P. Lubelski et al.9 performed a retrospective study to determine whether postoperative C5P can be predicted from preoperative antero-posterior diameter (APD), foraminal diameter (FD), and/or cord-lamina angle (CLA). 98 consecutive patients who underwent either anterior or posterior decompression surgery at C4-C5 for spondylotic myelopathy were analyzed. It was found that for every 1-mm increase in APD and FD, the odds of developing palsy decrease 69% (p<0.01) and decrease 98% (p<0.01), respectively. In contrast, for every 1-degree increase in CLA, the odds of developing palsy increase by 43% (p<0.01). Furthermore, Lubelski et al. used these three preoperative parameters - APD, FD, and CLA - to create a nomogram that predicts the probability that a patient will develop C5 palsy. This nomogram will be investigated for validity in the current study.

Preliminary Studies:

In addition to the study mentioned above, several authors have demonstrated the efficacy of prophylactic C5 foraminotomy during laminoplasty to prevent postoperative C5P. Sasai et al.7 performed the first prospective study using microcervical foraminotomy (MCF) during cervical laminoplasty as a prophylactic measure to prevent C5P. MCF was used selectively in patients with EMG abnormalities (Group A), and decreased the incidence of postoperative C5P compared to a group that did not have EMG studies or MCF performed (Group B). No patients in Group A and three patients in Group B experienced postoperative C5P (0% vs. 8.1%; p=0.035). No adverse outcomes were reported in this study. Based on these results, the authors suggested preexisting subclinical C5 root compression as a cause of C5P after posterior cervical decompression for myelopathy.

In 2012, Katsumi et al.5 performed a prospective, non-randomized study analyzing whether bilateral C5 foraminotomy can prevent C5P after open-door laminoplasty. Prophylactic bilateral foraminotomy done on 141 consecutive patients was seen to significantly decrease the incidence of postoperative C5P compared to a control group (1.4% and 6.4%, respectively; p<0.05). These results support the hypothesis that preoperative C5 foraminal stenosis is associated with a higher risk of C5P. Furthermore, these findings are consistent with the tethering phenomenon hypothesis regarding the pathomechanism of C5P. The only two patients in this study who developed C5P after undergoing prophylactic foraminotomy did not receive meticulous decompression of the C5 nerve root, leaving residual superior articular process. No patients in either group experienced postoperative infection or durotomy. Although the average operative time was longer in the foraminotomy group (102 minutes and 129 minutes, p<0.01), there was no significant difference in intraoperative blood loss between the two groups. In order to better elucidate the true effect of bilateral C5 foraminotomy, the procedure must be performed uniformly and randomized to all patients included.

With the current literature providing some evidence to suggest the efficacy of prophylactic bilateral C5 foraminotomies to reduce the incidence of postoperative C5P, there remains a need for a randomized, prospective study to investigate foraminotomy as a potentially beneficial procedure to all patients undergoing cervical decompression.

Significance of Proposed Study Bilateral foraminotomy has been correlated with a reduced risk of developing C5P following cervical decompression surgery, but an identical foraminotomy procedure has never been applied in a randomized manner to all qualifying patients in a study.5,6,7 Additionally, prophylactic foraminotomy has only been prospectively studied during laminoplasty. In the proposed study, bilateral foraminotomy will be randomized to patients receiving cervical decompression surgery (laminoplasty, laminectomy, fusion). Subsequently, incidence of C5P as well as other surgical complications will be monitored to determine efficacy of prophylactic C5 bilateral foraminotomy during cervical decompression.

Research Procedures:

This is a multicenter randomized trial, including the following sites: Cleveland Clinic, Columbia University Medical Center, and University of Southern California Spine Center. Patients undergoing cervical decompression surgery will be consented and enrolled if they meet the inclusion and exclusion criteria detailed above. The EPIC Electronic Medical Record database will be queried to retrieve medical records consistent with the study sample and to determine all cervical decompression surgeries. Patients' sex, race, date of birth, BMI, medical comorbidities, medications, history of spinal trauma or surgical intervention, smoking status/ history, spinal levels involved, type of surgery, operating surgeon, length of hospital stay, operative time, blood loss, in-hospital complications noted and patient complications following surgery will be obtained. Additionally, preoperative anteroposterior diameter of the spinal canal at C4-C5, ipsilateral foraminal diameter at C4-C5, and the morphological relationship between the spinal cord and the ipsilateral lamina (cord-lamina angle) will be obtained. Clinical outcome measures will be analyzed using standard statistical methods.

Intervention:

In addition to the decompression technique indicated directly for treatment of cervical myelopathy, bilateral keyhole foraminotomies will be done prophylactically in an attempt to minimize postoperative complications, specifically C5 Palsy. Under microscopic or loop magnification, a high-speed burr is used to perform the foraminotomy. The keyhole foraminotomy begins at the lamina-facet junction, with careful consideration of the amount of facet resection. Typically, only the medial one third is drilled. Then a 1- or 2-mm Kerrison punch can be carefully placed over the nerve root and then used to undercut the facet, ensuring that the spine is not destabilized by the foraminotomy. The amount of facet resection must not exceed 50% in order to preserve spine stability.

Consent:

All patients will be enrolled after completion of the attached informed consent form. All patients' information in this prospective study will be treated as confidential. This study involves no risk to the physician, or OR staff. A cervical foraminotomy is a common, short procedure (e.g. 5 minutes) that involves making more room for a cervical nerve root as it exits the spinal column. It is a procedure that all surgeons perform routinely, and in no way put the patient at risk for spine structural problems. Similarly, it does not impart additional measurable risk to the patient of neurological injury or infection over that risk already being incurred by the patient for the index procedure. Patients who are under the age of 18 will be excluded for previously mentioned scientific reasons. Women and minorities are expected to participate proportionally to their numbers diagnosed with cervical myelopathy.

ELIGIBILITY:
Inclusion Criteria:

* Cleveland Clinic patients who have been diagnosed with cervical myelopathy, without radiculopathy, and will undergo posterior cervical decompression involving the C4-C5 interspace between 2016 and 2018. This includes patients undergoing cervical laminoplasty and cervical laminectomy and fusion.

Exclusion Criteria:

* Any patient younger than 18 years of age will not be included on the basis of skeletal immaturity. Patients with C5 radiculopathy - defined in our study as the existence of preoperative deltoid muscle weakness in grade 3 or less by MMT - will be excluded. Any patients who have undergone previous cervical spine surgery, or who have any spinal malignancy, trauma or infection will be excluded in order to eliminate the confounding effect of multiple surgical interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
C5 Palsy | Upon discharge, 2 weeks postoperatively and 3 months postoperatively
  Using manual muscle testing and upper extremity sensory exam findings to determine C5 palsy status. C5P is defined as: a reduction of at least 1 in deltoid and/or biceps brachii manual muscle testing scores compared to preoperative scores, without any deterioration of myelopathic symptoms.

SECONDARY OUTCOMES:
Preoperative anatomic measurements | Preoperative
  Anteroposterior diameter, foraminal diameter and cord-lamina angle will be determined using preoperative computed tomography scan
Operative time | Intra-operative measurement
  Time length of operation
Blood loss | Intra-operative measurement
  Amount of blood loss during surgery
Back Pain | Preoperative, 2 weeks postoperative and 3 months postoperative
  Visual Analog Scale for Back Pain (0-10)
Leg Pain | Preoperative, 2 weeks postoperative and 3 months postoperative
  Visual Analog Scale for Leg Pain (0-10)
Emergency department visit | within 90 days postoperatively
  Subject has Emergency department visit
Readmission to hospital | within 90 days postoperatively
  Subject is readmitted to hospital within 90 days post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Mroz, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wada E, Suzuki S, Kanazawa A, Matsuoka T, Miyamoto S, Yonenobu K. Subtotal corpectomy versus laminoplasty for multilevel cervical spondylotic myelopathy: a long-term follow-up study over 10 years. Spine (Phila Pa 1976). 2001 Jul 1;26(13):1443-7; discussion 1448. doi: 10.1097/00007632-200107010-00011. PMID 11458148
- [Background] Elliott AY, Cleveland P, Cervenka J, Castro AE, Stein N, Hakala TR, Fraley EE. Characterization of a cell line from human transitional cell cancer of the urinary tract. J Natl Cancer Inst. 1974 Nov;53(5):1341-9. doi: 10.1093/jnci/53.5.1341. No abstract available. PMID 4431054
- [Background] Miller JA, Lubelski D, Alvin MD, Benzel EC, Mroz TE. C5 palsy after posterior cervical decompression and fusion: cost and quality-of-life implications. Spine J. 2014 Dec 1;14(12):2854-60. doi: 10.1016/j.spinee.2014.03.038. Epub 2014 Apr 3. PMID 24704502
- [Background] Sakaura H, Hosono N, Mukai Y, Ishii T, Yoshikawa H. C5 palsy after decompression surgery for cervical myelopathy: review of the literature. Spine (Phila Pa 1976). 2003 Nov 1;28(21):2447-51. doi: 10.1097/01.BRS.0000090833.96168.3F. PMID 14595162
- [Background] Katsumi K, Yamazaki A, Watanabe K, Ohashi M, Shoji H. Can prophylactic bilateral C4/C5 foraminotomy prevent postoperative C5 palsy after open-door laminoplasty?: a prospective study. Spine (Phila Pa 1976). 2012 Apr 20;37(9):748-54. doi: 10.1097/BRS.0b013e3182326957. PMID 21912316
- [Background] Komagata M, Nishiyama M, Endo K, Ikegami H, Tanaka S, Imakiire A. Prophylaxis of C5 palsy after cervical expansive laminoplasty by bilateral partial foraminotomy. Spine J. 2004 Nov-Dec;4(6):650-5. doi: 10.1016/j.spinee.2004.03.022. PMID 15541697
- [Background] Sasai K, Saito T, Akagi S, Kato I, Ohnari H, Iida H. Preventing C5 palsy after laminoplasty. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1972-7. doi: 10.1097/01.BRS.0000083237.94535.46. PMID 12973145
- [Background] Lubelski D, Derakhshan A, Nowacki AS, Wang JC, Steinmetz MP, Benzel EC, Mroz TE. Predicting C5 palsy via the use of preoperative anatomic measurements. Spine J. 2014 Sep 1;14(9):1895-901. doi: 10.1016/j.spinee.2013.10.038. Epub 2013 Nov 10. PMID 24225009